CLINICAL TRIAL: NCT03032159
Title: Text2Breathe: Enhance Parent Communication to Reduce Pediatric Asthma Disparities
Acronym: T2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: MultiCare Mary Bridge Children's Hospital & Health Center (Other)
Responsible Party: Principal Investigator, Tumaini Coker, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15488
Record Dates: First submitted 2016-04-20; First posted 2017-01-26 (Estimated); Results first posted 2024-11-01 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Participants randomized to the control group will receive their usual asthma care from their provider. Additionally, participants in the control group will receive reminder texts to schedule with their child's PCP and to get an annual flu shot. Participants will be surveyed over the phone for 20-30 minutes 3, 6, 12, 18, and 24 months after enrollment.
- Text2Breathe Study Group (Experimental): The "study" group spends about 10-20 minutes learning about ways to have better communication with their child's primary care provider about his/her asthma. Additionally this group is enrolled in the Text2Breathe messaging program which sends asthma related educational text messages 2 times a week for 3 months. Participants randomized to the study group will also receive reminder texts to schedule with their child's PCP and to get an annual flu shot. Participants will be surveyed over the phone for 20-30 minutes 3, 6, 12, 18, and 24 months after enrollment.
  Interventions: Behavioral: Text2Breathe Study Group

INTERVENTIONS:
Behavioral: Text2Breathe Study Group
  Arms: Text2Breathe Study Group

SUMMARY:
Text2Breathe (T2B) is a randomized controlled trial aimed at improving communication between parents and their children's' primary care providers about asthma. The overarching goal of this study is to reduce disparities among a population with high rates of pediatric asthma morbidity. The investigators are testing the efficacy of a short message service (SMS)-enhanced health communication (HC) intervention ("Text2Breathe") designed to equip urban, low-income parents with tools for communicating effectively with their children's primary care provider (PCP).

DETAILED DESCRIPTION:
Potentially eligible participants are approached and screened in person during an admission of their child to the emergency department for asthma care. Those participants randomized to the intervention will receive additional education on effective communication with their child's primary care provider (PCP). These participants will also receive educational text messages for three months after their initial visit. Text messages will include education on effectively communicating with their child's provider and general asthma information. Both the control group and intervention group will receive text message reminders to schedule regular follow up visits with their PCP and get an annual flu shot. Both groups will be contacted for follow up phone interviews at 3, 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Unlimited text messaging

Is the parent of child who is:

* Receiving asthma related care in the emergency department
* 2-12 years old inclusive
* Medicaid insured (no Private insurance)
* Physician diagnosed asthma for at least 12 months

Exclusion Criteria:

Is the parent of child who:

* Has seen a pulmonary or allergy sub-specialist more than once in the last 6 months
* Has seen a sub-specialist (not pulmonary or allergy) more than once in the last 12 months
* Has been hospitalized for more than 30 days
* Is currently enrolled in another asthma program or study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-08; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tumaini Coker, MD, MBA, Principal Investigator — Seattle Children's Hospital and Research Institute
Locations (2):
- United States (2):
  - Seattle Children's, Seattle, Washington
  - Mary Bridge Children's Hospital at Multi Care Health System, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (parents) were recruited from two children's hospitals in Seattle and Tacoma, Washington from 2015-2019.
Pre-assignment Details: Of the 661 potential parent participants screened for eligibility, 221 were eligible and randomized. Participants are unique parent/child dyads. The parents were enrolled, and each parent had a child that they provided data on. Those that were screened but excluded either did not meet inclusion criteria or declined to participate.
Groups:
- Control Group: Parents randomized to the control group child will receive their usual asthma care from their provider. Additionally, participants (parents) in the control group will receive reminder texts to schedule with their child's primary care provider (PCP) and to get an annual flu shot. Participants (parents) will be surveyed over the phone for 20-30 minutes 3, 6, 12, 18, and 24 months after enrollment.
- Text2Breathe Study Group: Parents in the "study" group spend about 10-20 minutes learning about ways to have better communication with their child's primary care provider about his/her asthma. Additionally, parents in this group were enrolled in the Text2Breathe messaging program which sends asthma related educational text messages 2 times a week for 3 months. Paret participants randomized to the study group will also receive reminder texts to schedule with their child's PCP and to get an annual flu shot. Parents will be surveyed over the phone for 20-30 minutes 3, 6, 12, 18, and 24 months after enrollment.
  Text2Breathe Study Group
Period: Overall Study
Arm/Group | Control Group | Text2Breathe Study Group
Started (Eligible parents randomized.) | 110 | 111
Completed (Completed 12-month Follow-Up Survey) | 91 | 77
Not Completed | 19 | 34

BASELINE CHARACTERISTICS:
Population: Parents enrolled into the control (usual care) group and intervention (Text2Breathe study group).
Groups:
- Control Group: Parents randomized to the control group child will receive their usual asthma care from their provider. Additionally, parents in the control group will receive reminder texts to schedule with their child's PCP and to get an annual flu shot. Parents will be surveyed over the phone for 20-30 minutes 3, 6, 12, 18, and 24 months after enrollment.
- Text2Breathe Study Group: Parents in the "study" group spend about 10-20 minutes learning about ways to have better communication with their child's primary care provider about his/her asthma. Additionally, parents in this group enrolled in the Text2Breathe messaging program which sends asthma related educational text messages 2 times a week for 3 months. Parents randomized to the study group will also receive reminder texts to schedule with their child's PCP and to get an annual flu shot. Parents will be surveyed over the phone for 20-30 minutes 3, 6, 12, 18, and 24 months after enrollment.
  Text2Breathe Study Group
- Total: Total of all reporting groups
Arm/Group | Control Group | Text2Breathe Study Group | Total
Number analyzed (Participants) | 110 | 111 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] — Child Age (years). Parents reported on age of child. We did not collect data on parent age
  years | 5.0 (2.3) | 6.4 (2.9) | 5.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Participant (Parent) reported sex
  Participants
    Female | 97 | 101 | 198
    Male | 13 | 10 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Parent race and ethnicity: Latino | 35 | 36 | 71
  Parent race and ethnicity: Non-Latino Black | 24 | 18 | 42
  Parent race and ethnicity: Multiracial | 2 | 12 | 14
  Parent race and ethnicity: Non-Latino White | 32 | 28 | 60
  Parent race and ethnicity: Other | 15 | 11 | 26
  Parent race and ethnicity: Missing | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 110 | 111 | 221

OUTCOME MEASURES:

1. Primary Outcome: Emergency Department Visits for Asthma Care
Description: Number of emergency department visits for asthma care
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ED visits
Groups:
- Text2Breathe Study Group: The "study" group spends about 10-20 minutes learning about ways to have better communication with their child's primary care provider about his/her asthma. Additionally this group is enrolled in the Text2Breathe messaging program which sends asthma related educational text messages 2 times a week for 3 months. Participants randomized to the study group will also receive reminder texts to schedule with their child's PCP and to get an annual flu shot. Participants will be surveyed over the phone for 20-30 minutes 3, 6, 12, 18, and 24 months after enrollment.
  Text2Breathe Study Group
Arm/Group | Control Group | Text2Breathe Study Group
Number analyzed (Participants) | 91 | 77
ED visits | 1.65 (1.7) | 1.95 (2.7)

2. Secondary Outcome: Asthma Morbidity
Description: Asthma morbidity measured as the number of days (or nights) of impairment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: max symptom days
Arm/Group | Control Group | Text2Breathe Study Group
Number analyzed (Participants) | 91 | 77
max symptom days | 3.36 (4.4) | 4.45 (5.0)

3. Other Pre Specified Outcome: Number of Scheduled Asthma Care Visits
Description: Number of visits with PCP for preventative asthma care in past 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Control Group | Text2Breathe Study Group
Number analyzed (Participants) | 91 | 77
number of visits | 2.07 (1.7) | 2.80 (3.0)

4. Other Pre Specified Outcome: Asthma Self-Management Questionnaire Standardized Score
Description: The Asthma Self-Management Questionnaire, recommended by experts convened for the Asthma Outcomes workshop, includes 16 multiple-choice questions regarding knowledge of preventive strategies and controller medication use. Standardized scores (0-100) are generated, with higher scores indicating more knowledge of self-management. Cronbach's alpha was 0.71. Wording of questions has been revised (e.g., "you" = "your child") to be appropriate for parents of children with asthma.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Text2Breathe Study Group
Number analyzed (Participants) | 91 | 77
score on a scale | 59.68 (17.2) | 58.67 (19.6)

5. Other Pre Specified Outcome: Parental Expectations for Child's Asthma Treatment Average Score
Description: In accordance with other research of pediatric asthma interventions, to assess parents' beliefs about possible asthma quality of life for their child we will administer an 8-item measure of parental expectations for asthma treatment. Parents respond to statements about their expectations (e.g., "I believe that my child can be symptom free most of the time.") using a 5-point Likert scale (1=strongly disagree to 5=strongly agree). Total scores are calculated by averaging across responses, and higher scores reflect more optimistic asthma outcome expectations (Cronbach's alpha = 0.70).
Time Frame: 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Parental Self-efficacy for Communicating With Healthcare Providers Self-competence Scale Summary Score
Description: The Medical Competence Communication Scale (MCCS) measures patient's perceptions of their own communication during their most recent medical visits. The patient version of the measure is used to assess information giving, seeking and verifying, as well as socio-emotional communication. The MCCS, patient version, consists of 23 items rated on a 5-point Likert scale (1= unimportant to 5= important) with a higher score indicating greater perception of communication competence (range 16-80). Cronbach's alpha ranges from 0.76-0.92 on the various subscales. Only the 16 self-competence items will be administered in this study. Wording of questions will be modified to state "my child's medical problem" rather than "my medical problem."
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Text2Breathe Study Group
Number analyzed (Participants) | 91 | 77
score on a scale | 78.72 (3.1) | 78.63 (3.1)

7. Other Pre Specified Outcome: Parental Asthma Management Self-efficacy Scale Summary Score
Description: The Parent Asthma Management Self-Efficacy Scale (PAMSES) is a valid and reliable instrument designed to measure parent self-efficacy in preventing and managing children's asthma attacks. The PAMSES consists of 13 items rated on a 5-point Likert scale (1=not at all sure to 5=completely sure) with a total possible score range of 13 to 65; higher scores indicate greater self-efficacy. Cronbach's alpha in a sample of primarily White mothers was 0.87.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the 12-month study period.
Description: Adverse events reported for the enrolled parent or their child.
Arm/Group | Control Group | Text2Breathe Study Group
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/111
Other Adverse Events (participants affected / at risk) | 0/110 | 0/111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT03032159/Prot_000.pdf
  • Statistical Analysis Plan (2014-07-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT03032159/SAP_001.pdf
  • Informed Consent Form (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT03032159/ICF_002.pdf